CLINICAL TRIAL: NCT04121013
Title: PREhospital Routage of Acute STroke Patients With Suspected Large Vessel Occlusion: Mothership Versus Drip and Ship, a Randomized Control Study in France (PRESTO-F)
Brief Title: PREhospital Routage of Acute STroke Patients With Suspected Large Vessel Occlusion: Mothership Versus Drip and Ship
Acronym: PRESTO-F
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2018-A02873-52
Record Dates: First submitted 2019-10-02; First posted 2019-10-09 (Actual); Last update posted 2021-04-14 (Actual); Status verified 2021-04

CONDITIONS: Stroke
Keywords: thrombectomy; drip'n'ship versus mothership; cost/effectiveness
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mothership (Active Comparator): Acute stroke patients with suspected large vessel occlusion will be directly transferred to the nearest transportation to the endovascular center
  Interventions: Other: mothership
- drip'n'ship (No Intervention): Acute stroke patients with suspected large vessel occlusion will be transferred to the closest local stroke centre or telemedicine hub as done with the current stroke protocol

INTERVENTIONS:
Other: mothership — Randomized controlled study: allocation to active or no intervention arm will be done accordingly to the design temporal sequence
  Arms: Mothership

SUMMARY:
Background: The outcome of ischemic stroke is related to the brain lesion volume and this volume of infarction is directly related to the time to reperfusion, which therefore depends on the time to initiation of therapy. Acute ischemic stroke is treated medically with the administration of intravenous rtPA, but recent randomized controlled trials have shown the efficacy of mechanical thrombectomy and is now the new gold standard in ischemic stroke. This new therapeutic strategy has created two possibilities for pre-hospital decision-making: i/ transport the patient directly to the nearest stroke unit to receive alteplase and then if indicated perform a thrombectomy (drip and ship) or ii/ bypassing thrombolysis centres in favour of endovascular thrombectomy (mothership).

Objective: To compare cost/effectiveness of transfer to the closest local stroke centre or telemedicine hub to direct transfer to the comprehensive stroke cent(CSC) in patients acute stroke with suspected large vessel occlusion.

Medical and economic expected impact: We hypothesize that direct transportation to CSC is associated with better clinical outcome in case of acute ischaemic stroke due to intracranial large vessel occlusion. However, we have to demonstrate that this approach is not associated with time from onset harm in patients not eligible to mechanical thrombectomy.

DETAILED DESCRIPTION:
Design: Multicenter, two-arm, prospective, open, blinded end-point (PROBE), randomized, clinical trial

Primary endpoint: Incremental cost-utility ratio at 12 months. Secondary endpoints: modified Rankin scale and EuroQoL5D scale at 3 months.

Eligibility criteria: A call to the emergency medical assistance service, 18 years and older, severe acute stroke symptoms, transportation time from scene to the CSC longer than time to go to the nearest stroke unit or telemedicine hub, transportation time from scene to the CSC compatible with IV thrombolysis, known time from onset, RACE score (assessed by medical emergency technicians) ≥5.

Experimental arm: direct transportation to the CSC. Control arm: transfer to the closest local stroke centre or telemedicine hub.

Sample size: 800 patients, 400 for each arm.

ELIGIBILITY:
Inclusion Criteria:

* A call to the emergency medical assistance service;
* age> 18y,
* known time of stroke onset;
* transportation time from scene to the CSC longer than time to go to the nearest stroke unit or telemedicine hub;
* transportation time from scene to the CSC compatible with IV thrombolysis;
* known time from onset, RACE score ≥5.

Exclusion Criteria:

* transportation time from scene to the CSC longer than time to go to the nearest stroke unit or telemedicine hub.
* no ambulance available
* bedridden patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2021-01-30 (Actual); Primary Completion 2022-01 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Incremental cost-utility ratio | 12 months
  Incremental cost-utility ratio (ICUR) at 12 months, defined as the ratio of the incremental cost of management by transfer to a CSC with MT (compared to the control arm "local PSC") to the gain in healthy survival (quality adjusted life years, QALYs).

SECONDARY OUTCOMES:
modified Rankin scale score | 90 days
  is a commonly used scale for measuring the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability. The scale runs from 0-6, running from perfect health without symptoms to death. Modified Rankin Scale score will be evaluated through a structured telephone-based interview performed by a central assessor who is blinded to group assignment

OTHER OUTCOMES:
EuroQoL5D scale | 90 days
  EQ-5D is a standardized instrument for measuring generic health status. In the description part, health status is measured in terms of five dimensions (5D); mobility, self-care, usual activities, pain/discomfort, and anxiety/depression.
  EuroQol5D scale will be evaluated through a structured telephone-based interview performed by a central assessor who is blinded to group assignment

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel Touze, Pr, Principal Investigator — University hospital of Caen
Locations (1):
- University hospital of Caen, Caen, Normanide, France

IPD SHARING:
Plan to Share IPD: No